CLINICAL TRIAL: NCT03236610
Title: Investigation of Efficacy of Tenofovir Monotherapy in Comparison With Entecavir Plus Tenofovir in Patients With Chronic Hepatitis B Patients Who Had Achieved Complete Viral Suppression on Entecavir Plus Tenofovir Combination Therapy-Multicenter Randomized Open-label Controlled Trial
Brief Title: Tenofovir Monotherapy in Patients With Chronic Hepatitis B Patients Who Had Achieved Complete Viral Suppression on Entecavir Plus Tenofovir
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uijeongbu St. Mary Hospital (Other)
Responsible Party: Principal Investigator, Chang Wook Kim, C.W. Kim, Uijeongbu St. Mary Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XC15MIMI0100U
Record Dates: First submitted 2017-07-28; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Proportion of Patients With a Sustained Virological Response (Serum HBV DNA <20 IU/mL) at Week 48
MeSH Terms: interventions — Tenofovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tenofovir (Experimental)
  Interventions: Drug: tenofovir monotherapy
- tenofovir plus entecavir (Active Comparator)
  Interventions: Drug: tenofovir plus entecavir combination

INTERVENTIONS:
Drug: tenofovir monotherapy — switching to tenofovir monotherapy
  Arms: tenofovir
Drug: tenofovir plus entecavir combination — continuing tenofovir plus entecavir
  Arms: tenofovir plus entecavir

SUMMARY:
Little is known about efficacy of switching to tenofovir monotherapy for multidrug-resistant chronic ehpatitis B patients who achieved a complete virological response to entecavir and tenofovir. This study aimed to investigate the efficacy of switching to tenofovir monotherapy for multidrug-resistant chronic hepatitis B patients with undetectable heaptitis B virus DNA while on tenofovir plus entecavir combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg (+) for > 6 months age >19 years antiviral resistance to LAM(rtL180M and/or M204V/I) & ADV (rtA181V/T and/or rtN236T) or ETV (rtT184A/C/F/G/I/L/S, rtS202G, or rtM250L/V, in addition to rtM204V/I) HBV DNA levels <20 IU/ml on two consecutive tests of 3-month interval currently receiving TDF+ETV for more than 12 months

Exclusion Criteria:

* Cr ≥1.5 mg/dL Evidence of decompensated liver disease Malignant neoplasm Coinfection with HIV, HCV

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
SVR at week 48 | 48 week
  Proportion of patients with a sustained virological response (serum HBV DNA <20 IU/mL) at week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Uijeongbu St. Mary Hospital, Uijongbu, South Korea